CLINICAL TRIAL: NCT06770608
Title: Comparison of Outcome of Microneedling With Autologous Platelet Rich Plasma Verses Microneedling With Topical Insulin in the Treatment of Post-Acne Atrophic Scars
Brief Title: Various Procedural Treatment Options for Post-acne Atrophic Scars
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Mohibullah Zahidi, Post Graduate Resident in Dermatology, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sheikh-ZMC
Record Dates: First submitted 2024-12-31; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Post-acne Atrophic Scars
Keywords: Microneedling; Autologous platelet rich plasma; Topical insulin; Post-acne atrophic scars

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micro-needling with topical human actrapid insulin group (Group A) (Active Comparator): Patients with post-acne atrophic scars will receive micro-needling with topical application of 2ml of human actrapid insulin
  Interventions: Procedure: micro-needling with topical human actrapid insulin
- Micro-needling with topical Platelet rich plasma(Group B) (Active Comparator): Patients with post-acne atrophic scars will receive micro-needling with topical application of 2ml Platelet rich plasma
  Interventions: Procedure: Micro-needling with topical Platelet rich plasma

INTERVENTIONS:
Procedure: micro-needling with topical human actrapid insulin — Micro-needling with topical application of 2ml of human actrapid insulin once monthly for 4 months
  Arms: Micro-needling with topical human actrapid insulin group (Group A)
Procedure: Micro-needling with topical Platelet rich plasma — Micro-needling with topical application of 2ml Platelet rich plasma once monthly for 4 months
  Arms: Micro-needling with topical Platelet rich plasma(Group B)

SUMMARY:
Post acne scars are formed as a result of very inflamed and nodulocystic acne. Most common type of acne scars are atrophic scars and they are further classified on the basis of depth and size of destruction into ice pick, boxcar and rolling scars. Evaulating the most efficacious, safe and affordable treatment option is the need of the hour. This study is going to compare the efficacy of microneedling with autologous platelet rich plasma verses microneedling with topical insulin in the treatment of post-acne atrophic scars as to find out the relatively more effective and safer treatment.

DETAILED DESCRIPTION:
Acne vulgaris is a disease involving inflammation or blockage of pilosebaceous units. Post acne scars are formed as a result of very inflamed and nodulocystic acne. There are many procedures to treat post-acne scar including lasers, platelet rich plasma, fillers, chemical peeling, pulsed dye lasers, fractional CO2 lasers, subcision and punch techniques, but almost lead to additional scaring and pigmentation.The major purpose of our study is comparison of outcome of micro-needling and platelet rich plasma as opposed to combining it with topical in atrophic scars due to acne, as topical insulin is natural component of body, cheap, easy to use, minimally invasive and a new therapy for post-acne scars. No local study was found in literature research. Hence, any effect of this potentially very effective therapeutic modality needs to be investigated.

OBJECTIVE: "To compare the outcome of microneedling with autologous platelet rich plasma verses microneedling with topical insulin in the treatment of post-acne atrophic scars".

Material & Methods: This randomized comarative study will be carried out in Outpatient Dermatology Department, Sheikh Zayed Hospital Rahim Yar Khan, Pakistan. Approval of the study has been taken from ethical review committee of the hospital.Data will be collected on prescribed form. Patient will be selected on basis of inclusion & exclusion criteria. Informed consent will be taken from selected patients before data collection. Study will includes 60 patients which will be divided into 2 groups A & B, 30 in each group. Group A will receive micro-needling with topical application of 2ml of human actrapid insulin. Group B will receive micro-needling with topical application of 2ml Platelet rich plasma. Face of the patient will be washed after 30 mints and patients will be strictly instructed regarding sun protection at least 1 day after the procedure. Blood glucose level will be checked prior to and 30 mints following procedure.

At monthly interval for total 4 sessions and follow up visit will be after 2 months of last session.Data will be analyzed by SPSS v25.0.

Chi-square test will be applied for qualitative variables and t-test will be used for quantitative variables.

ELIGIBILITY:
Inclusion Criteria:

* Age: 13-50 years
* Gender: both male and female
* Type of acne scar: Atrophic acne scar
* Patients not taking prior treatment in last 1-2 months

Exclusion Criteria:

* Pregnancy and lactating females
* Bleeding disorders
* Platelet count less than 100000
* Hypersensitivity to insulin, PRP
* Keloidal tendency
* Active herpes simples, warts and molluscum contagiosum
* Unrealistic expectations

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
To compare the outcome of microneedling with autologous platelet rich plasma verses microneedling with topical insulin in the treatment of post-acne atrophic scars | Clinical assessment for efficacy will be done monthly for 6 months
  Efficacy will be assesssed clinically at each follow up visit. Final efficacy of each treatment will be determined at last follow up visit( i.e. at 6th month after start of treatment).The final efficacy will be divided into following groups on the basis of clinical resolution of disease: 1.Remission: It is defined as complete resolution of all scar leaving behind normal skin. 2.Improvement: It is defined as a more than 50% healing of scars ,as clinically measured by the surface area from the baseline. 3.No improvement: It is defined as less than a 50% improvement in the healing of scars, as measured clinically by the surface area from the baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh zayed Medical College and Hospital, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No